CLINICAL TRIAL: NCT01536808
Title: Premature Aging and Type 2 Diabetes Mellitus: an Increased Risk of Cardiomyopathy?
Acronym: R2D2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008.506
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; accelerated aging; cellular senescence; diabetic cardiomyopathy; strain imaging; strain rate imaging,; echocardiography
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetic Cardiomyopathies | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Type 2 Diabetes Mellitus (Experimental)
  Interventions: Other: Cardiac RMI; Other: Analysis telomere; Other: Stress test; Other: echocardiography

INTERVENTIONS:
Other: Cardiac RMI — Cardiac RMI
Other: Analysis telomere — Analysis telomere
Other: Stress test — Stress test
Other: echocardiography — echocardiography

SUMMARY:
The potential clinical implications of this study are to optimise the selection of a population at risk for developing a diabetic cardiomyopathy among diabetic patients in order to develop early therapeutic strategies to prevent the left ventricular remodelling.

Therefore, the originality of this project is to hypothesize that :

* Diabetes mellitus is often associated with a premature aging syndrome
* Cellular senescence may potentiate the mechanisms that are involved in decreasing myocardial contractility in DM and,
* DM associated to premature aging may increase the risk of developing a cardiomyopathy Thus, the modulation of telomerase activity and the control of telomere length, together with the attenuation of the formation of reactive oxygen species, might represent important new targets in order to develop therapeutic tools in prevention of diabetic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus
* 40 < Age < 55 years old
* oral antidiabetic or insulin treatment
* No symptoms
* Sinus rhythm
* no sign or history of heart disease
* LVEF > 55%
* Absence of regional left ventricular motion abnormalities.

Exclusion Criteria:

* absence of sinus rhythm,
* silent ischemia defined as positive exercise test or positive stress echocardiography,
* history of cardiomyopathy or CAD,
* valvular heart disease hemodynamically significant,
* severe renal insufficiency defined as creatinine clearance < 30 mL/min,
* echocardiographic images unsuitable for quantification,
* type 1 diabetes mellitus,
* Important diabetes mellitus imbalance defined as glycated hemoglobin > 9% or glycemia > 3g/L uncontrolled hypertension (> 180/100 mmHg).

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Telomere shortening | 36 months
  Investigate whether biomarkers for senescence determined from blood samples, including telomere shortening and telomerase activity in diabetic patients have an impact of left ventricular remodelling as compared with age-matched controls and biological aged control subjects.

SECONDARY OUTCOMES:
Dysfunction by speckle tracking imaging | 36 months
  Study the incidence of subtle regional myocardial dysfunction by speckle tracking imaging (longitudinal and radial systolic strain)
Determine the predictive value of alteration | 36 months
  Determine the predictive value of alteration : Proteinuria, glycosylated haemoglobin, diabetes mellitus duration, blood pressure, BNP dosage, MRI diagnoses
Cardiovascular events | 36 months
  Investigate the predictive value of all those factors( telomere shortening, telomerase activity, echo abnormalities) on cardiovascular events including MI, HF, arrhythmia; ACV

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Dérumeaux, MD, Principal Investigator — Hospices Civils de Lyon - Hôpital Louis Pradel
Locations (1):
- Laboratoire d'échocardiographie, Bron, France

REFERENCES:
- [Background] Sen I, Trzaskalski NA, Hsiao YT, Liu PP, Shimizu I, Derumeaux GA. Aging at the Crossroads of Organ Interactions: Implications for the Heart. Circ Res. 2025 May 23;136(11):1286-1305. doi: 10.1161/CIRCRESAHA.125.325637. Epub 2025 May 22. PMID 40403108